CLINICAL TRIAL: NCT00275457
Title: A Randomised, Double-blind, Placebo-controlled Dose Titration Trial With 0.125-0.75 mg Pramipexole (Sifrol®) Orally to Investigate the Safety and Efficacy in Out-patients With Idiopathic Restless Legs Syndrome for 6 Weeks Followed by 46 Weeks Open-label or Double-blind Treatment Period
Brief Title: Efficacy and Safety of Pramipexole (PPX) in Moderate to Severe Idiopathic Restless Legs Syndrome (RLS) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 248.520
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: pramipexole

SUMMARY:
To evaluate safety and efficacy of pramipexole in the treatment of patients suffering from moderate to severe RLS over 6 weeks under double blinded conditions followed by a 46 week open label or double blind extension.

DETAILED DESCRIPTION:
To evaluate safety and efficacy of pramipexole in the treatment of patients suffering from moderate to severe RLS over 6 weeks under double blinded conditions followed by a 46 weeks open label or double blind extension

Study Hypotheses:

Null hypothesis: No difference between pramipexole and placebo in RLSRS total score from baseline and no difference in the CGI-I responder rates at the end of the 6 weeks double-blind treatment.

Comparison(s):

Pramipexole vs. Placebo

ELIGIBILITY:
Inclusion criteria:

1. Male or female out-patients aged 18-80
2. Diagnosis of idiopathic RLS according to the Clinical RLS criteria of the International RLS Study Group. All of the four criteria must be present:

   * Irresistible urge to move usually associated with sensory complaints of the lower limbs
   * Motor restlessness
   * Worsening of the symptoms at rest with at least partial and temporary relief by activity
   * Increased severity in the evening or at night
3. RLS rating scale for severity score > 15
4. RLS symptoms present at least 2 to 3 days per week within in the last 3 months
5. Written informed consent consistent with ICH/GCP and local legislation given prior to any study procedures
6. Ability and willingness to comply with study treatment regimen and to attend study assessments

Exclusion criteria:

1. Women of childbearing potential, who do not use adequate protection such as barrier protection, intrauterine device, or hormonal (oral or subcutaneous) contraception or postmenopausal women less than 6 months after last menses, surgically sterilised, oophorectomised or hysterectomised less than 3 months after operation and not using adequate protection or women neither using adequate protection nor being postmenopausal and their partner is not sterilised at least 6 months post operation or does not use condom, or any women not having negative serum pregnancy test at screening
2. Males not using an adequate form of contraception (condom, sterilisation at least 6 months post operation)
3. Patients who are breastfeeding
4. Concomitant or previous pharmacologically therapy of RLS as follows:

   * Any intake of levodopa within 5 days prior to baseline visit (V2)
   * Any intake of dopamine agonists within 14 days prior to baseline visit (V2)
   * History of any intake of pramipexole
5. Current (less than 14 days before treatment with trial medication or concomitant) treatment with medication or dietary supplements, which could significantly influence RLS symptoms - withdrawal symptoms caused by stopping any of the drugs above
6. Confirmed diagnose of diabetes mellitus requiring insulin therapy
7. Clinically significant renal disease or creatinine higher than upper limit of normal (ULN) at screening
8. Clinically significant hepatic disease or sGPT > 2 times the upper limit of normal range at screening
9. Clinical or laboratory signs of microcytic anaemia at the investigators discretion
10. Any of the following lab results at screening:

    * Hb or erythrocyte count below lower limit of normal (LLN)
    * Basal TSH, T3 or T4 clinically significantly (at the investigator's discretion) out of normal range at screening (if not caused by substitution therapy according the investigator's opinion)
11. Other clinically significant metabolic-endocrine, haematological, gastro-intestinal disease or pulmonary disease. Poorly controlled cardiovascular disease
12. History or clinical signs of peripheral neuropathy (PNP) of any origin in physical, neurological examination, myelopathy or multiple sclerosis or any other neurological disease, with potential to secondarily cause RLS symptoms
13. Presence of any other sleep disorder, such as, REM sleep behaviour disorder, narcolepsy or sleep apnoea syndrome
14. History of Schizophrenia or any psychotic disorder, history of mental disorders due to a general medical condition or any present axis I psychiatric disorder according DSM IV requiring any medical therapy or history of or alcohol abuse or drug addiction within the last 2 years before screening
15. Participation in a drug study within two months prior to the start of this study
16. History of or clinical signs for any form of epilepsy or seizures apart from fever related seizures in early childhood
17. History of or clinical signs of malign neoplasm
18. Patients on a shift-work-schedule, or who are otherwise unable to follow a regular sleep-wake cycle enabling use of study medication at times indicated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346
Dates: Start 2002-10; Primary Completion 2004-04 (Actual); Study Completion 2004-04

PRIMARY OUTCOMES:
Mean change from baseline to week 6 on the RLSRS +
CGI-I responders (much and very much improved)

SECONDARY OUTCOMES:
RLRS responders, CGI, PGI responders, EPSS, QoL (SF-36) VAS severity of RLS

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (33):
- Austria (7):
  - Univ.-Klinik für Neurologie, Graz
  - Univ.-Klinik für Neurologie, Innsbruck
  - AKH der Stadt Linz, Linz
  - Confraternität Privatklinik, Vienna
  - AKH Universitätsklinik für Psychiatrie, Vienna
  - Sonderkrankenanstalt für neurologischen und, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
- Germany (8):
  - Boehringer Ingelheim Investigational Site, Bad Dürrheim-Sunthausen
  - Boehringer Ingelheim Investigational Site, Bad Krozingen
  - Boehringer Ingelheim Investigational Site, Berlin
  - emovis GmbH, Berlin
  - Facharzt für Neurologie, Emmendingen
  - Boehringer Ingelheim Investigational Site, Kehl
  - ClinPharm International GmbH & Co. KG, Leipzig
  - Universitätsklinikum Giessen und Marburg, Marburg
- Netherlands (8):
  - Boehringer Ingelheim Investigational Site, Beek en Donk
  - Boehringer Ingelheim Investigational Site, Deurne
  - Boehringer Ingelheim Investigational Site, Ewijk
  - Boehringer Ingelheim Investigational Site, Lichtenvoorde
  - Boehringer Ingelheim Investigational Site, Rijswijk
  - Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - Boehringer Ingelheim Investigational Site, Rotterdam
  - Boehringer Ingelheim Investigational Site, The Hague
- Norway (3):
  - Boehringer Ingelheim Investigational Site, Hamar
  - Boehringer Ingelheim Investigational Site, Oslo
  - Boehringer Ingelheim Investigational Site, Tønsberg
- Sweden (7):
  - Boehringer Ingelheim Investigational Site, Gothenburg
  - Boehringer Ingelheim Investigational Site, Örebro
  - Stockholms Neuro Center, Stockholm
  - Neurologkliniken, Stockholm
  - Boehringer Ingelheim Investigational Site, Uppsala
  - Läkarhuset Vällingby, Vällingby
  - Boehringer Ingelheim Investigational Site, Västra Frölunda